CLINICAL TRIAL: NCT05687149
Title: Defining the Natural History of Squamous Cell Carcinoma in Fanconi Anemia
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001109; 001109-C
Record Dates: First submitted 2023-01-14; First posted 2023-01-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12-23

CONDITIONS: Fanconi Anemia; Inherited Bone Marrow Failure Syndrome
Keywords: Hereditary; Inherited Bone Marrow Failure Syndrome; Oral Potentially Malignant Lesion; Surveillance; Precancer
MeSH Terms: conditions — Fanconi Anemia; Congenital Bone Marrow Failure Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fanconi anemia: A prospective cohort of individuals with Fanconi anemia (FA) at very high risk of squamous cell carcinoma (SCC)

SUMMARY:
Background:

Fanconi anemia (FA) is an inherited disorder. People with FA are more likely to get certain cancers, especially squamous cell carcinoma (SCC). These cancers usually appear first in the mouth, esophagus, and genital and anal areas. Early detection of SCCs may help improve survival rates for people with FA.

Objective:

This natural history study will regularly screen people with FA for SCC.

Eligibility:

People aged 12 years and older with FA or a prior cancer diagnosis. Children aged 8 to 11 years with FA may also be eligible.

Design:

Participants will receive a comprehensive screening for cancer or early signs of cancer.

Participants will have a physical exam. They will provide blood and saliva samples. Cells will be collected by rubbing a swab on the inside of the cheeks. A skin sample may be removed from the back, buttocks, or inside of the upper arm.

Participants will have pictures taken of their mouth. Any mouth sores will be mapped. Cells will be collected from the sores with a small brush.

Specialists will examine the participant s ears, nose, throat, teeth, and skin.

Adult participants may have a gastrointestinal exam or pelvic exam. Participants may have an endoscopy. A long tube with a camera and a light will be inserted through the mouth and down into the stomach.

Participants may have a liver ultrasound. A wand will be pressed against their belly to get pictures of the organs inside the body.

Participants will have screenings every year for up to 10 years. Each visit will last up to 3 days. They will have remote follow-up visits every 6 - 8 months....

DETAILED DESCRIPTION:
Study Description:

This is a natural history study involving questionnaires, clinical and research evaluations, clinical and research laboratory tests, review of medical records, and cancer surveillance. A prospective cohort of individuals with Fanconi anemia (FA) at very high risk of squamous cell carcinoma (SCC) will be screened and provide new information on oral potentially malignant lesion (OPML) development and robustly quantify the risk of progression of OPML to cancer in FA.

Objectives:

Primary Objectives:

1. To establish a central program and a team of expert clinicians and scientists at the NIH Clinical Center to conduct a comprehensive longitudinal study of cancer screening in adolescent and young adults (AYA) with FA at high risk of SCC through detailed clinical evaluation and biospecimen collection.
2. To characterize the clinical and pathological natural history of OPMLs in AYAs with FA using brush biopsies for cytopathologic diagnosis and DNA aneuploidy and correlate those findings with tissue biopsies and genomic analyses of oral epithelial dysplasia (OED) and SCC.
3. To prospectively screen individuals with FA for early indicators for the development of esophageal and anogenital SCC and hematological malignancy.

Secondary Objectives:

1. To identify genetic, epigenetic, and immunologic mechanisms underlying tumorigenesis and immune escape in individuals with FA.
2. To facilitate the enrollment of individuals with FA with high-grade dysplasia or SCC in intra- and extra-mural precision intervention trials.

Endpoints:

Primary Endpoints:

1. Characterize the natural history of OPMLs in FA, rates of progression, regression, and development of new lesions
2. Determine the utility of brush biopsy to identify oral dysplasia and SCC in FA
3. Identify potential precursor states for esophageal and anogenital cancers in FA
4. Develop screening guidelines for esophageal and anogenital cancer in FA

Secondary Endpoints:

1. Identify predictive biomarkers of oral SCC development
2. Characterize genetic and epigenetic changes that lead to SCC development
3. Facilitate patient enrollment in intervention trials

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. On referral, persons >= 12 years with FA primarily from North America will be included. An individual with FA who is 8 - 11 years can also be included if they have a history of persistent OPMLs, dysphagia, or other concerning symptoms.
  2. Individuals with prior cancer diagnosis are eligible.
  3. Individuals from other countries are eligible provided they can travel to the USA on their own.
  4. Ability to understand and/or the willingness of the individual, parent, LAR, or minor s legal guardian to provide informed consent.

EXCLUSION CRITERIA:

1. Referred individuals for whom reported diagnosis of FA cannot be verified.
2. Inability of the individual, parent, LAR, or legal guardian to understand and be willing to sign a written informed consent document.

Ages: 8 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons >=12 years with FA primarily from North America will be included in the study. Persons < 12 years can also be included if they have a history of persistent oral potentially malignant lesions, dysphagia, or other concerning symptoms. Persons with FA from other countries are eligible provided they can travel to USA on their own.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Screen Patients with FA | ongoing
  Prospectively screen individuals with FA for early indicators for the development of esophageal and anogenital SCC.
Clinical and Pathological Natural History of Oral Potentially Malignant Lesion | ongoing
  Characterize the clinical and pathological natural history of OPMLs in AYAs with FA using brush biopsies for cytopathologic diagnosis and aneuploidy and correlate those findings with tissue biopsies and genomic analyses of oral epithelial dysplasia (OED) and SCC.
Cohort of Patients with FA | ongoing
  A prospective cohort of individuals with Fanconi anemia (FA) at very high risk of squamous cell carcinoma (SCC)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J McReynolds, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Velleuer E, Dietrich R, Pomjanski N, de Santana Almeida Araujo IK, Silva de Araujo BE, Sroka I, Biesterfeld S, Bocking A, Schramm M. Diagnostic accuracy of brush biopsy-based cytology for the early detection of oral cancer and precursors in Fanconi anemia. Cancer Cytopathol. 2020 Jun;128(6):403-413. doi: 10.1002/cncy.22249. Epub 2020 Feb 5. PMID 32022466
- [Background] Alter BP, Giri N, Savage SA, Rosenberg PS. Cancer in the National Cancer Institute inherited bone marrow failure syndrome cohort after fifteen years of follow-up. Haematologica. 2018 Jan;103(1):30-39. doi: 10.3324/haematol.2017.178111. Epub 2017 Oct 19. PMID 29051281
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001109-C.html